CLINICAL TRIAL: NCT01238315
Title: A Phase Ib Study of the Safety and Preliminary Efficacy of Allogeneic Intracerebral Human Central Nervous System Stem Cell Transplantation in Subjects With Non-Refractory Infantile and Late Infantile Neuronal Ceroid Lipofuscinosis
Brief Title: Safety and Efficacy Study of HuCNS-SC in Subjects With Neuronal Ceroid Lipofuscinosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of timely patient accrual
Sponsor: StemCells, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-N03-NCL
Record Dates: First submitted 2010-11-05; First posted 2010-11-10 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Neuronal Ceroid Lipofuscinosis
Keywords: Batten's disease; INCL; LINCL; Neuronal Ceroid Lipofuscinosis; NCL
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HuCNS-SC (Other)
  Interventions: Biological: HuCNS-SC

INTERVENTIONS:
Biological: HuCNS-SC — Surgery to implant human CNS stem cells
  Other Names: human neural stem cells; stem cells; neural stem cells

SUMMARY:
The purpose of this Phase Ib study is to determine if "Human Central Nervous System Stem Cells"(HuCNS-SC) is safe to be transplanted in subjects with infantile and late infantile neuronal ceroid lipofuscinosis. The study will also measure post-transplantation disease progression.

DETAILED DESCRIPTION:
Participation in this study will involve screening assessments, surgery to implant HuCNS-SC, medication to suppress immune system and a series of follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 6 years
* Male or female
* Clinical diagnosis of Infantile neuronal ceroid lipofuscinosis or late infantile neuronal ceroid lipofuscinosis
* CLN1 or CLN2 mutation

Exclusion Criteria:

* Previously received an organ, tissue or bone marrow transplantation
* Previously participated in any gene or cell therapy study
* Infection with hepatitis virus, cytomegalovirus, Epstein-Barr virus, or Human Immunodeficiency Virus (HIV)
* Current or prior cancer
* Bleeding disorder
* Unable to have an MRI scan

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
number of participants with adverse events. | one year following transplantation
  Safety will be measured by number of adverse events and changes in neurological status.

SECONDARY OUTCOMES:
Number of subjects with improvement in neurological, neuropsychological development, MRI and MRS | one year following transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Selden, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- See also: Related Info — http://www.stemcellsinc.com